CLINICAL TRIAL: NCT05144451
Title: Transcranial Doppler and Neurological Complications After Liver Transplantation
Brief Title: Transcranial Doppler During Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MD.21.09.535
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Liver Transplantation; Ultrasonography, Doppler, Transcranial; Complication, Postoperative; Neurologic Deficits
MeSH Terms: conditions — Postoperative Complications; Neurologic Manifestations | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: A single-arm trial involving 100 patients undergoing living donor liver transplantation; all will be examined using transcranial doppler to find out its predictive value on post-transplant neurological deficits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCD arm (Experimental): All patients will be evaluated with TCD for prediction of the post-transplant neurological complications
  Interventions: Diagnostic Test: Transcranial Doppler

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler — Transcranial Doppler-derived parameters; pulsatility index (PI), resistance index (RI), mean flow velocity (Vmean) will be recorded before induction of anesthesia (T1).
  After induction, TCD parameters, Hemodynamic variables including heart rate (HR), invasive mean arterial blood pressure (MAP), and central venous pressure (CVP) together with Arterial blood gases (ABG analysis with values of PH, PCO2, PO2, blood oxygen saturation SO2 and bicarbonate HCO3), end-tidal carbon dioxide (ETCO2) and body temperature will be recorded too. Just before skin incision (T2), at the end of anhepatic phase 5 minutes before reperfusion (T3), 5 minutes after reperfusion (T4) and at the end of surgery (T5).
  Postoperatively at ICU, TCD parameters, Hemodynamic variables, and ABG will be obtained 24 hours postoperative (T6) and at discharge from ICU (T7).
  Other Names: TCD

SUMMARY:
This is a prospective study that would investigate the transcranial doppler (TCD) changes during the living donor liver transplantation and the association between the TCD changes and the post-transplant neurological complications.

DETAILED DESCRIPTION:
Objectives:

Participants & Setting:

Intervention & Measurements:

Sample size:

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for living donor liver transplantation for whatever the indication at Gastrointestinal surgery center (GISC)

Exclusion Criteria:

* Patients with coexisting neuropsychiatric or cerebrovascular disorders or those who have a history of head trauma or brain surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-11-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Post-transplant Neurological Complication | 28 days after transplantation
  incidence of Neurological Complication as a composite outcome (tremors, seizures, demyelination, posterior reversible encephalopathy syndrome, stroke)

SECONDARY OUTCOMES:
flow patterns throughout the transplant surgery and in the ICU | intraoperative and 7 days after transplantion
  normal, hyperemic, low-flow, or vasospastic flow by TCD

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, MD, Study Director — Mansoura University Faculty of Medicine
Locations (1):
- Mansoura University, Gastrointestinal Surgery Center, Liver Transplantation Unit, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available with the corresponding author at reasonable request. The Data publishing with the manuscript will be discussed later.
Time Frame: will be updated
Access Criteria: will be updated